CLINICAL TRIAL: NCT04875520
Title: Assessing Testing Strategies for Safe Return to K-12 Schools in an Underserved Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202104013
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-02

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Screening testing; School-based COVID-19 Transmission
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Screening testing plus symptomatic testing (Active Comparator): Among 16 middle and high schools, 8 will be randomized to offer students and staff weekly SARS-CoV-2 testing. Additionally, these schools will offer testing for symptomatic students, staff, household members in all age groups.
  Interventions: Other: Screening testing strategy
- Symptomatic testing (Active Comparator): All 16 schools will have testing available for individuals that have symptoms or need a test for other reasons.
  Interventions: Other: No screening testing strategy

INTERVENTIONS:
Other: Screening testing strategy — The intervention we are evaluating is the use of weekly screening testing among students and staff.
  Arms: Weekly Screening testing plus symptomatic testing
Other: No screening testing strategy — a group of schools will not receive screening testing.
  Arms: Symptomatic testing

SUMMARY:
The primary goal of this study is to determine the most effective SARS-CoV-2 testing strategy for successful return of in-person school in the under-served communities of St. Louis.

Regular screening testing has been recommended by the CDC as an additive mitigation strategy for in-person schools in areas of high community transmission. We will compare the effectiveness and acceptance of two different school-based testing strategies among students and school staff (symptomatic testing only versus weekly surveillance testing plus symptomatic testing), measuring school-based SARS-CoV-2 transmission through a cluster randomized trial.

DETAILED DESCRIPTION:
We will complete a cluster randomized trial to compare the incidence of school-based SARS-CoV-2 transmission between weekly screening testing of students and school staff versus testing only symptomatic students and staff. In this proposal, 16 middle and high schools from five school districts in the St. Louis metropolitan area will be cluster randomized to screening testing plus symptomatic testing versus symptomatic testing alone. The symptomatic testing will be provided to the entire school community as well as household members of students and staff.

The second Aim will evaluate existing mitigation strategies utilized in schools and the rate of school-based SARS-CoV-2 transmission by defining the mitigation strategies utilized in participating schools through survey tools developed with CDC and their impact on school-based COVID-19 transmission and quantifying the rate of COVID-19 transmission in schools and the impact of this transmission on households through extensive interviews and testing of contacts and household members.

Our 3rd Aim involves partnering with community-based organizations to specify and address the social, ethical, and behavioral implications of in-person schooling during the COVID-19 pandemic and the impact of SARS-CoV-2 testing on the school and community. Listening sessions will be utilized to understand barriers and facilitators to testing, ethical concerns of the community in research participation, and the behavioral health impact of lack of in-person schooling.

ELIGIBILITY:
Inclusion Criteria:

* A student or staff in one of the five school districts.
* Household members of a student or staff member in the five school districts.

Exclusion Criteria:

* People not affiliated with the school.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1390 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason G. Newland, MD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Ferguson-Florissant School District, Hazelwood, Missouri
  - Jennings School District, Jennings, Missouri
  - Pattonville School District, Saint Ann, Missouri
  - Normandy Schools Collaborative, St Louis, Missouri
  - The School District of University City, University City, Missouri

REFERENCES:
- [Background] Van Dyke ME, Mendoza MCB, Li W, Parker EM, Belay B, Davis EM, Quint JJ, Penman-Aguilar A, Clarke KEN. Racial and Ethnic Disparities in COVID-19 Incidence by Age, Sex, and Period Among Persons Aged <25 Years - 16 U.S. Jurisdictions, January 1-December 31, 2020. MMWR Morb Mortal Wkly Rep. 2021 Mar 19;70(11):382-388. doi: 10.15585/mmwr.mm7011e1. PMID 33735165
- [Background] Bryant DJ, Oo M, Damian AJ. The rise of adverse childhood experiences during the COVID-19 pandemic. Psychol Trauma. 2020 Aug;12(S1):S193-S194. doi: 10.1037/tra0000711. Epub 2020 Jun 18. PMID 32551773
- [Background] Benner AD, Mistry RS. Child Development During the COVID-19 Pandemic Through a Life Course Theory Lens. Child Dev Perspect. 2020 Dec;14(4):236-243. doi: 10.1111/cdep.12387. Epub 2020 Oct 15. PMID 33230400
- [Background] Zimmerman KO, Akinboyo IC, Brookhart MA, Boutzoukas AE, McGann KA, Smith MJ, Maradiaga Panayotti G, Armstrong SC, Bristow H, Parker D, Zadrozny S, Weber DJ, Benjamin DK Jr; ABC SCIENCE COLLABORATIVE. Incidence and Secondary Transmission of SARS-CoV-2 Infections in Schools. Pediatrics. 2021 Apr;147(4):e2020048090. doi: 10.1542/peds.2020-048090. Epub 2021 Jan 8. PMID 33419869
- [Background] Falk A, Benda A, Falk P, Steffen S, Wallace Z, Hoeg TB. COVID-19 Cases and Transmission in 17 K-12 Schools - Wood County, Wisconsin, August 31-November 29, 2020. MMWR Morb Mortal Wkly Rep. 2021 Jan 29;70(4):136-140. doi: 10.15585/mmwr.mm7004e3. PMID 33507890
- [Background] Orscheln RC, Newland JG, Rosen DA. Practical School Algorithms for Symptomatic or SARS-CoV-2-Exposed Students Are Essential for Returning Children to In-Person Learning. J Pediatr. 2021 Feb;229:275-277. doi: 10.1016/j.jpeds.2020.09.060. Epub 2020 Sep 25. No abstract available. PMID 32980377
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Lalli MA, Langmade SJ, Chen X, Fronick CC, Sawyer CS, Burcea LC, Wilkinson MN, Fulton RS, Heinz M, Buchser WJ, Head RD, Mitra RD, Milbrandt J. Rapid and extraction-free detection of SARS-CoV-2 from saliva with colorimetric LAMP. medRxiv [Preprint]. 2020 Aug 6:2020.05.07.20093542. doi: 10.1101/2020.05.07.20093542. PMID 32511508
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Derived] Hayes S, Malone S, Bonty B, Mueller N, Reyes SM, Reyes SA, Evans C, Wilcher-Roberts M, Watterson T, Akuse S, Shelley J, Yuan G, Lackey I, Prater J, Montgomery B, Williams C, Butler-Barnes ST, Harris K, Caburnay C, Dougherty NL, Liu J, Lai A, Neidich J, Fritz S, Newland JG. Assessing COVID-19 testing strategies in K-12 schools in underserved populations: study protocol for a cluster-randomized trial. BMC Public Health. 2022 Jun 13;22(1):1177. doi: 10.1186/s12889-022-13577-z. PMID 35698094
- See also: Johnson A, Buford T. Early Data Shows African Americans Have Contracted and Died of Coronavirus at an Alarming Rate. Propublica. 2020. Accessed March 11, 2021 — http://www.propublica.org/article/early-data-shows-african-americans-have-contracted-and-died-of-coronavirus-at-an-alarming-rate
- See also: Henderson MB, West MR, Peterson PE. Pandemic Parent Survey Finds Perverse Pattern: Students are More Likely to Be Attending School in Person Where COVID Is Spreading More Rapidly. Education Next. 2021;21(2). Accessed March 11, 2021 — https://www.educationnext.org/pandemic-parent-survey-finds-perverse-pattern-students-more-likely-to-be-attending-school-in-person-where-covid-is-spreading-more-rapidly

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All students, staff, and family members from 16 middle and high schools were eligible to participate.
Pre-assignment Details: 1390 individuals from 16 middle and high schools were enrolled.
Units Other Than Participants: schools
Period: Overall Study
Arm/Group | Weekly Screening Testing Plus Symptomatic Testing | Symptomatic Testing
Started | 894; 8 schools | 496; 8 schools
Completed | 797; 8 schools | 460; 8 schools
Not Completed | 97; 0 schools | 36; 0 schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Screening Testing Plus Symptomatic Testing | Symptomatic Testing | Total
Number analyzed (Participants) | 894 | 496 | 1390
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [16 to 47] | 30 [13 to 48] | 35 [15 to 47]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 530 | 299 | 829
  Gender: Male | 310 | 175 | 485
  Gender: Other | 54 | 22 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 7 | 37
  Not Hispanic or Latino | 771 | 413 | 1184
  Unknown or Not Reported | 93 | 76 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 9 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 323 | 282 | 605
  White | 431 | 144 | 575
  More than one race | 47 | 31 | 78
  Unknown or Not Reported | 79 | 36 | 115
Participant Type [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 843 | 469 | 1312
    Staff | 353 | 203 | 556
    Student | 200 | 183 | 383
    Household | 290 | 83 | 373
Received COVID-19 Vaccine [Count of Participants; unit: Participants] — Other = prefer not to answer and unknown.
  Participants
    Yes | 509 | 252 | 761
    No | 170 | 142 | 312
    Other | 215 | 102 | 317
Social Vulnerability Index [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 875 | 491 | 1366
    Low | 293 | 120 | 413
    Low-Medium | 128 | 67 | 195
    Medium - High | 331 | 197 | 528
    High | 123 | 107 | 230

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of All COVID-19 Cases in Schools.
Description: The rate of all new COVID-19 cases of student/staff in schools per randomization group.
Time Frame: Up to one year.
Population: The unit analyzed were the number of the tests completed overall during the study.
Measure: Count of Units; unit: Completed tests
Units Other Than Participants: Completed tests
Groups:
- Weekly Screening Testing Plus Symptomatic Testing; Symptomatic Testing: Total reported school cases during study period divided by school population.
Arm/Group | Weekly Screening Testing Plus Symptomatic Testing | Symptomatic Testing
Number analyzed (Participants) | 894 | 496
Number analyzed (Completed tests) | 6436 | 7488
Completed tests | 453 | 297
Statistical Analysis 1: Comparison: Weekly Screening Testing Plus Symptomatic Testing vs Symptomatic Testing; Test type: Non-Inferiority — Overall rate compared using GEE model includes any person affiliated with the school who tested positive at least once during the study period that the schools reported to us that were positive. This includes people in our testing program and not in our testing program; p = 0.25, generalized estimating equations; Mean Difference (Final Values) = -0.01845, 95% CI 2-sided [-0.04981 to 0.01292]

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and non-serious adverse events were not assessed for study participants.
Arm/Group | Weekly Screening Testing Plus Symptomatic Testing | Symptomatic Testing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size. Local and federal COVID-19 recommendations and precautions were continuously changing. The omicron surge in St. Louis presented an unforeseeable strain on the study's testing resources, and symptomatic testing had to be paused for 37 days. Due to the specific PCR test utilized not being designed for a high positivity rate. Study experienced lower recruitment than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04875520/Prot_SAP_000.pdf